CLINICAL TRIAL: NCT00385476
Title: Cancer Patients' Medication Knowledge in the Emergency Center
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2003-0526
Record Dates: First submitted 2006-10-05; First posted 2006-10-09 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Medication Knowledge; Emergency Center; Questionnaire; Survey

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient Medication Knowledge Tool: Assessment of Cancer patients' knowledge of their medications in an outpatient acute care setting
  Interventions: Behavioral: PMKT Questionnaire

INTERVENTIONS:
Behavioral: PMKT Questionnaire — Patient Medication Knowledge Tool - Questionnaire entailing the medications the patient is currently taking.

SUMMARY:
The goal of the study is to learn about patients' knowledge of their medications in an outpatient acute care setting (such as the M. D. Anderson Emergency Center) and to learn about any clinical factors that affect patients' knowledge of their medications.

DETAILED DESCRIPTION:
You will be asked to list your prescription medicines, over-the-counter medicines, herbal preparations and vitamins, minerals and supplements that you take. Information about you (such as age or gender), the status of the disease (such as cancer diagnosis and extent of disease), and your Emergency Center visit (such as your reason for visit and discharge diagnosis) will be collected from your medical record.

To find out if your answers on the questionnaire are correct regarding the medications you take, researchers will check the pharmacy database for medications you fill at the M. D. Anderson pharmacy, your medical record, and contact any outside pharmacy that you may use to fill your medicines, with your permission. In order for outside pharmacies to release the requested medication information, you will need to sign an Authorization for Disclosure of Health Information from Pharmacy Records.

Your information will be kept confidential. All patient data will be reported and published as a group. You will not be individually identified. Data will be stored with patient codes so that your identity will be protected. In addition, the study database will be password protected.

You may be contacted in the future for more information; however, you are not obligated to answer any future questions just because you agreed to participate in this study.

This is an investigational study. About 350 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to the Emergency Center
2. Patients must be able to read and write English
3. Patients must agree to participate and sign informed consent
4. Patients 16 years or above. (Age limit explained below)
5. Patients must be able to complete the survey tool. They may have help from a caregiver in transcribing the information but the caregiver can not fill the tool independent of the patient. A research assistant will be trained to discriminate whether a caregiver is acting as a scriber or independently completing the tool. If the caregiver completes the tool independently, the patient will be excluded from the study.

Exclusion Criteria:

1. Patients with altered mental status and those with an acute, emergent illness and hemodynamic instability (Examples: status epileptics, sepsis, and cardiac arrest)
2. Employees of the institution with work-related injuries
3. Visitors who are non-cancer patients
4. Patients transferred directly from another hospital
5. Patients will be excluded after their first enrollment during the study period. (Can only be enrolled once though may have multiple Emergency Center visits during study time frame).
6. Patients will be excluded if all prescribed medications are filled at an external pharmacy and this pharmacy is not accessible.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants admitted to the UT MD Anderson Cancer Center Emergency Center.
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2005-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Patients' knowledge of their medications in an outpatient acute care setting (such as the M. D. Anderson Emergency Center). | 4 Years

SECONDARY OUTCOMES:
Results of the Patient Medication Knowledge Tool (Questionnaire) | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Escalante, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org